CLINICAL TRIAL: NCT00305201
Title: Cardiovascular Risk Markers Before and After Therapy With Statins in Patients With History of Kawasaki Disease
Brief Title: Cardiovascular Risk Markers and Response to Statins After Kawasaki Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn due to lack of study participants
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Arturo Borzutzky, MD, Pontificia Universidad Catolica de Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PG-29/05
Record Dates: First submitted 2006-03-20; First posted 2006-03-21 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Kawasaki Disease
Keywords: Mucocutaneous Lymph Node Syndrome; Kawasaki disease; Endothelial dysfunction; Pravastatin; Statin therapy
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome | interventions — Pravastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: pravastatin

SUMMARY:
The purpose of this study is to determine whether Chilean children with history of Kawasaki disease have endothelial dysfunction years after the acute phase of the disease, and if this condition can be modified by treatment with statins.

DETAILED DESCRIPTION:
Kawasaki disease (KD) in its acute phase produces endothelial inflammation that can lead to dilatation and aneurysms of coronary and peripheral arteries. This initial injury leads to persistent endothelial dysfunction several years after having the disease. As a consequence, these patients may have a higher cardiovascular risk than general population. Studies with HMG-CoA reductase inhibitors (statins) have suggested that these have an anti-inflammatory effect over the endothelium, that may be independent of its lipid-lowering effects. The hypothesis of this study is that KD produces endothelial dysfunction that is persistent years after acute disease, and that this dysfunction can be modified by treatment with statins.The study consists of two phases. On the first we will perform ultrasound assessment of endothelial-dependent flow-mediated vasodilation of the brachial artery and evaluate other cardiovascular risk markers in patients and healthy controls. On the second phase patients with history of Kawasaki disease will be randomized and allocated to treatment with Pravastatin or placebo, after which a new evaluation of flow-mediated dilation of the brachial artery and cardiovascular risk markers will be performed.

Comparison(s): Children older than 8 years of age with history of Kawasaki disease more than 12 months before enrollment, compared with paired by age children without history of KD or other cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* History of Kawasaki disease more than 12 months before enrollment
* Present age of 8 years or older

Exclusion Criteria:

* Diabetes mellitus
* Not controlled hypertension
* Treatment with drugs thay modify endothelial function such as angiotensin converting enzyme inhibitors, angiotensin II receptor antagonists, and calcium channel blockers
* Smokers of more than 5 cigarettes per day
* Total cholesterol higher than 250 mg/dl
* Triglycerides higher than 300mg/dl
* Chronic treatment with statins
* Chronic renal insufficiency (creatinine > 1.5 mg/dl)

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2006-04; Study Completion 2007-05 (Estimated)

PRIMARY OUTCOMES:
Percent of change in brachial artery dilatation after statin therapy

SECONDARY OUTCOMES:
Decrease in LDL
Increase in HDL
Decrease in triglycerides
Decrease in high sensitivity CRP

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Borzutzky, MD, Principal Investigator — Pontificia Universidad Catolica de Chile, School of Medicine, Department of Pediatrics; Miguel Gutierrez, MD, Study Director — Pontificia Universidad Catolica de Chile, School of Medicine, Department of Rheumatology and Clinical Immunology
Locations (1):
- Pontificia Universidad Catolica de Chile, School of Medicine, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Background] Kato H, Sugimura T, Akagi T, Sato N, Hashino K, Maeno Y, Kazue T, Eto G, Yamakawa R. Long-term consequences of Kawasaki disease. A 10- to 21-year follow-up study of 594 patients. Circulation. 1996 Sep 15;94(6):1379-85. doi: 10.1161/01.cir.94.6.1379. PMID 8822996
- [Background] Dhillon R, Clarkson P, Donald AE, Powe AJ, Nash M, Novelli V, Dillon MJ, Deanfield JE. Endothelial dysfunction late after Kawasaki disease. Circulation. 1996 Nov 1;94(9):2103-6. doi: 10.1161/01.cir.94.9.2103. PMID 8901658
- [Background] Furuyama H, Odagawa Y, Katoh C, Iwado Y, Ito Y, Noriyasu K, Mabuchi M, Yoshinaga K, Kuge Y, Kobayashi K, Tamaki N. Altered myocardial flow reserve and endothelial function late after Kawasaki disease. J Pediatr. 2003 Feb;142(2):149-54. doi: 10.1067/mpd.2003.46. PMID 12584536
- [Background] de Jongh S, Lilien MR, op't Roodt J, Stroes ES, Bakker HD, Kastelein JJ. Early statin therapy restores endothelial function in children with familial hypercholesterolemia. J Am Coll Cardiol. 2002 Dec 18;40(12):2117-21. doi: 10.1016/s0735-1097(02)02593-7. PMID 12505222